CLINICAL TRIAL: NCT06596005
Title: A Randomized, Double-blind, Placebo Parallel-controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of TJ0113 Capsule in Patients With Early-stage Parkinson's Disease
Brief Title: Efficacy and Safety of TJ0113 Capsule in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Taizhou Hospital (Other); Wenzhou Central Hospital (Other); Sir Run Run Shaw Hospital (Other); The Second Affiliated Hospital of Jiaxing University (Other); Hangzhou PhecdaMed Co., Ltd. (Industry); Huzhou Central Hospital (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TJJS01-201
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Results first posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TJ0113 200mg (Experimental): Subjects will receive 200 mg of TJ0113 capsules for 12 consecutive weeks
  Interventions: Drug: TJ0113 200mg
- TJ0113 400mg (Experimental): Subjects will receive 400 mg of TJ0113 capsules for 12 consecutive weeks
  Interventions: Drug: TJ0113 400mg
- Placebo (Placebo Comparator): Subjects will receive 200 mg or 400 mg of placebo for 12 consecutive weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TJ0113 200mg — 200 mg Capsule, Once Daily
  Arms: TJ0113 200mg
Drug: TJ0113 400mg — 400 mg Capsule, Once Daily
  Arms: TJ0113 400mg
Drug: Placebo — Capsule, Once Daily
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo parallel-controlled Phase II clinical trial to evaluate the efficacy and safety of TJ0113 capsule in patients with early-stage Parkinson's disease

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo parallel-controlled phase II clinical trial which is designed to assess the efficacy and safety of TJ0113 capsules in the treatment of patients with early-stage Parkinson's disease (PD). It is planned to include approximately 150 subjects with early-stage PD who will be randomized in a 1: 1 ratio into two cohorts (Cohort 1: 200 mg dose group; Cohort 2: 400 mg dose group). Within each cohort, subjects who have been successfully screened will be randomly assigned to TJ0113 capsule group and the placebo group in a ratio of 2: 1 within each stratum based on a stratification factor whether they have been receiving levodopa, the background medication for PD (yes vs. no) at a stable dose. Among them, approximately 50 subjects will receive TJ0113 capsules and approximately 25 subjects will receive the placebo. In this study, there will be approximately 50 subjects in each of the TJ0113 capsules 200 mg group, TJ0113 capsules 400 mg group and the placebo group.

After randomization, subjects will receive the oral administration of TJ0113 capsules or the placebo for 12 consecutive weeks and continue to receive follow-up visits for 1 week after the end of treatment. For subjects who have been receiving the anti-PD drug at a stable dose for at least 4 weeks prior to study entry, the original regimen of the background medication for PD should be maintained during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily participate in the clinical trial, and have signed the informed consent form (ICF), are able to understand and follow the study protocol, willing to visit the study site on time, fully understand the content, process and potential adverse reactions of the study, and indicate the date of signing the ICF;
2. Males or females aged 30-80 years (both inclusive) at the time of signing the ICF;
3. Subjects who are diagnosed with PD according to the Diagnostic Criteria for Parkinson's Disease in China (2016 edition);
4. The scores of modified Hoehn and Yahr Scale at screening are 1-2.5 (both inclusive);
5. Subjects who have not previously received anti-PD drugs; or those who have previously used any anti-PD drugs but have not received such drug within 4 weeks before study entry; or those who have received the anti-PD drug at a stable dose for at least 4 weeks before study entry and agree to maintain the original treatment regimen during the study;
6. Subjects with the scores of MDS-UPDRS Part III of ≥ 22 at screening (it should be scored ≥ 12 hours apart from the most recent dose of the anti-PD drug for subjects who have been receiving an anti-PD drug at a stable dose for at least 4 weeks prior to study entry);
7. Subjects of childbearing potential (including spouses of male subjects) who have no childbearing or sperm donation plan from the end of the screening period to within 6 months after the last dose and are willing to use at least one effective method (see Appendix I for details) for contraception.

Exclusion Criteria:

1. Presence of any medical condition that may interfere with full participation in the study, including but not limited to the following: medical history of epilepsy or any complications, medical history of hemolytic anemia, pulmonary embolism, respiratory depression, active psychiatric disease, or malignancy;
2. Subjects who have experienced a New York Heart Association (NYHA) Class III or above congestive heart failure, unstable angina pectoris, acute myocardial infarction, hemorrhagic stroke (stroke), and ischemic stroke (including transient ischemic attack) within 6 months before screening; or those who have undergone any percutaneous coronary intervention or coronary artery bypass grafting, heart valve repair/replacement; or those with severe arrhythmia as judged by the investigator at the time of screening;
3. Subjects with prior personal or family history of long-QT syndrome, family history of sudden death of any immediate family members (meaning a parent, child, or sibling) prior to the age of 40 years; and/or personal history of unexplained syncope within 1 year prior to screening; and/or QTcF > 450 ms (male), QTcF > 470 ms (female) measured by Electrocardiogram(ECG) at rest during screening;
4. Subjects with unstably controlled hypertension at screening, defined as the systolic blood pressure ≥ 160 mmHg and/or the diastolic blood pressure ≥ 100 mmHg (verify before randomization);
5. Subjects with symptomatic orthostatic hypotension at screening, or who experiences a decrease in systolic blood pressure of ≥ 30 mmHg or a decrease in diastolic blood pressure of ≥ 15 mmHg within 3 minutes when changing from the supine to the standing position (verify before randomization);
6. Atypical PD (e.g., Parkinsonism, multiple system atrophy, progressive supranuclear palsy), or secondary PD (e.g., delayed or drug-induced PD);
7. Subjects who have clinically significant hepatic insufficiency which is defined as the total bilirubin (TBIL) &amp;gt; 2 × upper limit of normal (ULN) or alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) &amp;gt; 2 × ULN;
8. Subjects who have clinically significant renal insufficiency (creatinine clearance [Ccr] &amp;lt; 30 mL/min, see the calculation formula in Appendix II);
9. Any condition (e.g., severe arthritis, severe dyskinesia, traumatic injury with permanent physical disability) that may affect the MDS-UPDRS motor examination;
10. Subjects who have a history of suicidal intention (including actual attempts, interrupted attempts, or failed attempts) and are at risk of committing suicide as judged by the investigator;
11. Subjects who suffer from severe mental abnormalities (anxiety, depression) as judged by the investigator, and the depression or anxiety score as rated by the Part I of the MDS-UPDRS is ≥ 3 at screening;
12. Subjects who have taken any serotonin reuptake inhibitors (such as fluoxetine, paroxetine, trazodone, citalopram, escitalopram, etc.) within 4 weeks prior to screening;
13. Subjects who have dementia or moderate or above cognitive dysfunction and the MDS-UPDRS score for 1.1 cognitive impairment is ≥ 3 at screening;
14. Subjects who have a history of surgical treatment for PD (e.g., deep brain stimulation, pallidotomy, etc.), or those who have undergone any major or medium surgery or have experienced any serious trauma or serious infection within 3 months prior to screening, those who are unsuitable for this study at the discretion of the investigator or plan to undergo any surgical treatment (excluding an outpatient surgery that has no impact on subject safety or study results as judged by the investigator) during the study;
15. Subjects who have participated in a clinical trial that involves the administration of an investigational drug (a new chemical entity), device, or surgery within 3 months or 5 half-lives before screening, whichever is longer;
16. Subjects with evidence of alcoholism (≥ 14 units of alcohol per week on average, 1 unit ≈ 360 mL of beer, 45 mL of liquor, or 150 mL of wine) or drug abuse within 6 months prior to screening that may interfere with the subject&amp;#39;s understanding of the study or completion of the study as judged by the investigator;
17. Subjects who are known to have hypersensitivity/allergic reaction or intolerance to any component of the investigational product;
18. Positive for any of the hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, and Treponema pallidum antibody (TP-Ab) at screening;
19. Pregnant or breastfeeding women;
20. Subjects who are unable to swallow oral drugs, or have any condition that may significantly affect the absorption, distribution, metabolism and excretion of the drug, or any condition that may pose a hazard to subjects participating in the study, as judged by the investigator;
21. Subjects who have a history of organ transplantation (excluding corneal transplantation);
22. Subjects who have donated or lost blood of ≥400 mL, or received blood transfusions within 3 months prior to screening;
23. Subjects who have any other conditions that may affect study compliance as deemed by the investigator, or those who are unable to participate in the study for their own reasons.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Luo, Doctor, Principal Investigator — Sceond Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TJ0113 200mg | TJ0113 400mg | Placebo
Started | 50 | 48 | 51
Completed | 48 | 44 | 50
Not Completed | 2 | 4 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Other | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TJ0113 200mg | TJ0113 400mg | Placebo | Total
Number analyzed (Participants) | 50 | 48 | 51 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (7.93) | 59.9 (7.90) | 60.3 (10.02) | 60.0 (8.64)
Age, Customized [Count of Participants; unit: Participants]
  <18 | 0 | 0 | 0 | 0
  18-65 | 35 | 38 | 32 | 105
  66-75 | 15 | 10 | 17 | 42
  >75 | 0 | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 19 | 65
  Male | 29 | 23 | 32 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 50 | 48 | 51 | 149
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 50 | 48 | 51 | 149
MDS-UPDRS Score at Baseline(Part III) [Mean (Standard Deviation); unit: units on a scale] — The Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) rating tool was used to follow longitudinal course of Parkinson's Disease. It was made up of 4 parts.
  In this study, the Part III score was designated as the primary efficacy endpoint.Part 3: Motor examination (18 items, some of which include multiple scorable components, resulting in a total of 33 scoreable entries, with an overall score ranging from 0 to 132).Higher values represent a worse outcome.
  units on a scale | 47 (9.93) | 46.8 (10.60) | 45.1 (9.69) | 46.3 (10.04)

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in Scores of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III (Motor Examination) in Subjects After 12 Weeks of Treatment.Evaluation Time Point: ≥ 12 Hours From the Most Recent Dose of Anti-PD Drug.
Description: The Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) rating tool was used to follow longitudinal course of Parkinson's Disease. It was made up of 4 parts.
  In this study, the Part III score was designated as the primary efficacy endpoint.Part 3: Motor examination (18 items, some of which include multiple scorable components, resulting in a total of 33 scoreable entries, with an overall score ranging from 0 to 132).Higher values represent a worse outcome.
Time Frame: After 12 weeks.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | TJ0113 200mg | TJ0113 400mg | Placebo
Number analyzed (Participants) | 50 | 48 | 51
score on a scale | -7.06 (0.703) | -7.40 (0.714) | -0.69 (0.686)
Statistical Analysis 1: Comparison: TJ0113 200mg vs Placebo; Test type: Other; p < 0.0001, MMRM — The LSM, SE, and difference from placebo with 95% CI and nominal P-value are estimated using MMRM, with baseline MDS-UPDRS Part III scores and L-Dopa use as covariates, and treatment group, visit, and group-by-visit interaction as fixed effects; Difference in least squares means = -6.37, 95% CI 2-sided [-8.09 to -4.64], Standard Error of Mean 0.871
Statistical Analysis 2: Comparison: TJ0113 400mg vs Placebo; Test type: Other; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in least squares means = -6.70, 95% CI 2-sided [-8.45 to -4.95], Standard Error of Mean 0.886

ADVERSE EVENTS:
Time Frame: AEs are collected in this trial from the time the subject receives the investigational product (i.e., TJ0113 capsules or placebo) until the end of the follow-up period.(From enrollment to end of treatment at 13 weeks.)
Arm/Group | TJ0113 200mg | TJ0113 400mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/48 | 0/51
Serious Adverse Events (participants affected / at risk) | 2/50 | 0/48 | 0/51
Other Adverse Events (participants affected / at risk) | 25/50 | 28/48 | 25/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TJ0113 200mg (N=50) | TJ0113 400mg (N=48) | Placebo (N=51)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TJ0113 200mg (N=50) | TJ0113 400mg (N=48) | Placebo (N=51)
White blood cell count decreased (Investigations) | 2 (2) | 2 (2) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (2) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 2 (3)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Bile acids increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Urinary occult blood positive (Investigations) | 0 (0) | 0 (0) | 2 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram ST segment depression (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 1 (2) | 0 (0)
Interleukin level increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Periodontitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Rapid eye movements sleep abnormal (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-02-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT06596005/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-22): https://cdn.clinicaltrials.gov/large-docs/05/NCT06596005/SAP_001.pdf